CLINICAL TRIAL: NCT05940558
Title: A Phase IIa, Open Label, Single-centre Study to Assess the Initial Antifibrotic Efficacy, Safety, Tolerability, Pharmacokinetic and Pharmacodynamic Profile of MBF-118 in Crohn's Disease Patients with Stenosis
Brief Title: Safety and Efficacy of MBF-118 in Patients with Crohn Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Medibiofarma S.L. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MBF-118CT-02
Record Dates: First submitted 2023-06-29; First posted 2023-07-11 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MBF-118 100mg oral multiple dose (Experimental): Drug: MBF-118 100mg oral capsules. Single daily dose. One hard gelatin capsules during 28 days.
  Subjects who have previously completed 28 days treatment with 100 mg MBF-118 and did not show any serious adverse effects will have the option to participate to a 90-day treatment.
  Interventions: Drug: MBF-118 oral capsules
- MBF-118 200mg oral multiple dose (Experimental): Drug: MBF-118 100mg oral capsules. Single daily dose. Two hard gelatin capsules during 28 days
  Interventions: Drug: MBF-118 oral capsules

INTERVENTIONS:
Drug: MBF-118 oral capsules — MBF-118 oral capsules PPAR gamma receptor partial agonist

SUMMARY:
This is a Phase IIa (proof of concept), single center clinical trial to evaluate the safety and efficacy of daily MBF-118 oral treatment during 28 days in Crohn's disease patients on top of standard of care.

DETAILED DESCRIPTION:
This is a Phase 2a study to evaluate the safety, tolerability and exploratory efficacy of daily oral treatment with either 100 mg or 200 mg MBF-118 during 28 days in Crohn's disease patients diagnosed with stenosis, in order to provide reliable safety, tolerability, and PK data that will guide drug dose and therapeutic regimen choices in subsequent clinical studies.

The study design is a single-center, open-label group consisting of two cohorts, one dosed with 100 mg MBF-118 daily for 28 days and one dosed with 200 mg MBF-118 daily for 28 days, in approximately 5 subjects per cohort without placebo control. No randomisation is required. The first five patients to start initiate the trial will be dosed with 100 mg. The subsequent five patients initiating the trial will be dosed with 200 mg.

For each subject, the study duration will last a total of approximately 14-16 weeks consisting of a screening period of 2-4 weeks, a treatment period of 4 weeks and a follow-up period of 8 weeks.

The subjects who have previously completed 28 days treatment with 100 mg MBF-118 and did not show any serious adverse effects will have the option to participate to an open-label 90-day extension phase. The extension phase will last approximately 19-21 weeks consisting of up to 21 days screening, 90 treatment days and 42 follow-up days.

ELIGIBILITY:
Inclusion Criteria:

* Participants must meet each of the following criteria for enrolment into the study:

  1. Male or nonpregnant, nonlactating females, age 18-75. Males and females of childbearing potential must agree to use adequate birth control measures during the study. Females of childbearing potential must have a negative serum pregnancy test prior to Visit 2 and either be sexually abstinent or must use a hormonal (oral, implantable, or injectable) or double barrier method of birth control throughout the study, and until 60 days after the last dose of study drug. Females unable to bear children must have documentation of such in the source records (i.e., tubal ligation, hysterectomy, or postmenopausal [defined as a minimum of 1 year since the last menstrual period]).
  2. Diagnosis of CD based on clinical, endoscopic, and histologic evidence established at least 3 months prior to Screening.
  3. Has mild to severe ileal and/or colonic CD.
  4. Participant has no more than 4 naïve or anastomotic small bowel strictures by MRE or IU in the terminal ileum at Screening. A stricture is defined as:

     1. localized luminal narrowing (luminal ≤ 50% relative to normal adjacent bowel); AND
     2. wall thickening (≥ 125% relative to adjacent bowel); AND
     3. length < 20 cm
  5. If participants are using a treatment for CD, they should be on a stable dose for at least 3 months prior to study commencement. Acceptable treatments include non-steroidal anti-inflammatory drugs (NSAIDs) and anti-inflammatory biologics.
  6. Ability to participate fully in all aspects of this clinical trial. Full comprehension of consent language and written informed consent must be obtained from the participant and documented.

Exclusion Criteria:

Participants who exhibit any of the following conditions are to be excluded from the study:

1. CD-related complications:

   * Previous ileorectal anastomosis, or a proctocolectomy. Patients who have received colonic resection are allowed in this study.
   * Short bowel syndrome
   * Ileostomy, colostomy, small bowel stoma, or ileoanal pouch
   * Fistulae in or adjacent to an ileal stenosis. Participants with perianal fistulae could be included if not septic. Participants with internally penetrating fistulae are excluded.
   * Suspected or diagnosed active intra-abdominal or perianal abscess that has not been appropriately treated
   * Toxic megacolon
2. Use of corticosteroid treatment for symptoms of inflammatory bowel disease within the last 2 weeks. Corticosteroids should not be taken during the screening, treatment or follow-up periods of the trial.
3. History or current diagnosis of ulcerative colitis, indeterminate colitis, ischemic colitis, nonsteroidal anti-inflammatory drug (NSAID)-induced colitis, idiopathic colitis (i.e., colitis not consistent with CD), radiation colitis, microscopic colitis, colonic mucosal dysplasia, or untreated bile acid malabsorption.
4. Uncontrolled primary sclerosing cholangitis.
5. Malignancies or history of malignancy within 5 years of the initial screening visit (V1), except for adequately treated or completely excised non-metastatic basal cell carcinoma, squamous cell carcinoma of the skin, or cervical carcinoma in situ.
6. Has a severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration, or may interfere with the interpretation of study results, as determined by the investigator.
7. Patients with cardiac failure or history of cardiac failure (New York Heart Association (NYHA) stages I to IV congestive heart failure) and patients with prior myocardial infarction or symptomatic coronary artery disease.
8. Clinically significant abnormal clinical laboratory values, vital signs, physical examination, or 12-lead electrocardiogram (ECG) at Screening or Baseline [PR ≥ 220 msec, QRS ≥120 msec and QTc ≥ 440 msec, bradycardia (<50 bpm) or clinically significant minor ST wave changes or any other abnormal changes on the screening ECG that would interfere with measurement of the QT interval].
9. Systemic or opportunistic infections including:

   * Patients with active tuberculosis (TB) determined at Screening, defined as a positive QuantiFERON test, or a purified protein derivative (PPD) skin test. Patients who test positive and show symptoms of TB (abnormal chest x-ray, or positive sputum smear or culture, active TB bacteria in his/her body, usually feels sick and may have symptoms such as coughing, fever, and weight loss) will be excluded. Patients positive for TB who develop symptoms during the study period will be removed from the trial. An exception is made for subjects with a history of latent TB who are currently receiving treatment for latent TB, will initiate treatment for latent TB before the first dose of study treatment, or have documentation of completing appropriate treatment for latent TB within 3 years prior to the first dose of study treatment). Patients who test positive for TB during the study period but who do not show symptoms will be allowed to continue the study.
   * Active infection with HIV.
   * Evidence of positive hepatitis B surface antigen (HBsAg) or hepatitis B core antibody (HBcAb). NOTE: if a participant tests negative for HBsAg, but positive for HBcAb, the participant would be considered eligible if no presence of HBV DNA is confirmed by HBV DNA polymerase chain reaction reflex testing performed in the central laboratory.
   * Chronic hepatitis C (HCV) (positive HCVAb and HCV RNA). Note: Participants who are HCVAb positive without evidence of HCV RNA may be considered eligible (spontaneous viral clearance or previously treated and cured).
   * Evidence of Clostridioides difficile toxin or treatment for C. difficile infection, or other intestinal bacterial pathogen, within 30 days prior to Screening.
   * History of invasive fungal infections such as Candida or Aspergillus within 6 months prior to randomization.
   * History of herpes (simplex type 1, simplex type 2, or zoster) infection or reactivation within 12 weeks prior to randomization, or frequent recurrence of herpes (more than 2 times per year).
   * Evidence of active cytomegalovirus (CMV) infection at Screening.
   * Any other clinically significant extraintestinal infection or opportunistic, chronic, or recurring infection within 6 months before Screening. Examples include, but are not limited to, infections requiring intravenous (IV) antibiotics, hospitalization, or prolonged treatment.
10. Concurrent or previous participation in another clinical trial and received investigational therapy within 4 weeks or 5 half-lives (whichever is longer) prior to Screening. Fecal microbiota transplant (includes human microbiota-based therapeutics) within 4 weeks prior to Screening are allowed.
11. Any major surgery, in the investigator's opinion, performed within 8 weeks prior to randomization or planned during the study (i.e., any surgical procedure requiring general anesthesia).
12. Unwillingness to withhold protocol-prohibited medications during the trial.
13. History of excessive alcohol or drug abuse that, in the opinion of the investigator, may interfere with the participant's ability to comply with the study procedures.
14. Known or suspected allergy, anaphylaxis, hypersensitivity or intolerance to the study drug(s) or its' excipients.
15. Prior enrolment in the current study and had received study treatment.
16. The participant is an immediate family member, study site employee, or is in a dependent relationship with a study site employee who is involved in conduct of this study (e.g., spouse, parent, child, sibling).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-09-10 (Actual); Study Completion 2024-09-10 (Actual)

PRIMARY OUTCOMES:
Number of Adverse events | 12 weeks
  Evaluate the safety of MBF-118 administered for 28 days in subjects with Crohn's disease by assessing the number, severity, and type of adverse events.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela, Galicia, Spain

IPD SHARING:
Plan to Share IPD: No